CLINICAL TRIAL: NCT05740527
Title: Ambulatory Closed-loop Stimulation to Inhibit Neurogenic Bladder Over-activity
Brief Title: Ambulatory Closed-loop Stimulation for Bladder Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MetroHealth Medical Center (Other)
Collaborators: The Craig H. Neilsen Foundation (Other)
Responsible Party: Principal Investigator, Dennis Bourbeau, Principal Investigator, MetroHealth Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-00690
Record Dates: First submitted 2023-02-01; First posted 2023-02-23 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: Urinary Bladder, Neurogenic
Keywords: spinal cord injury; bladder; urinary incontinence; stimulation; closed loop; reducing bladder spasms
MeSH Terms: conditions — Urinary Bladder, Neurogenic; Spinal Cord Injuries; Urinary Incontinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Testing closed-loop system in an ambulatory setting (Other): Closed-loop system feasibility testing
  Interventions: Device: Noninvasive electrical stimulation of genital nerves

INTERVENTIONS:
Device: Noninvasive electrical stimulation of genital nerves — A closed-loop system (in-bladder sensor, radio, algorithm, and stimulator) is being tested for the feasibility of inhibiting neurogenic bladder overactivity in an ambulatory setting.

SUMMARY:
Individuals with spinal cord injury (SCI) develop neurogenic detrusor overactivity (NDO), resulting in urinary incontinence, decreased bladder capacity, and reduced quality of life. Current treatments incompletely address the problem and have unwanted side effects. Therefore, an alternative approach is needed. Electrical stimulation of the genital nerves (GNS) can inhibit NDO, improving bladder capacity and urinary continence. However, an automated closed-loop bladder feedback system, which currently does not exist, is necessary for individuals with SCI and NDO to utilize this therapy. The researchers have developed a custom algorithm to detect bladder contractions in real time, which requires only a bladder pressure signal. Our collaborators have developed a wireless, catheter-free bladder pressure sensor, called the UroMonitor, that was recently approved for testing in human participants. The goal of this project is to evaluate the potential feasibility and effectiveness of automated closed-loop GNS to inhibit unwanted bladder contractions using our custom algorithm and the wireless UroMonitor sensor. This project represents the next logical step toward improving or restoring bladder control using existing or emerging approaches to meet an important need for individuals with SCI. Successful completion of this project will motivate advancing a closed-loop approach using our custom algorithm and wireless bladder pressure sensor.

DETAILED DESCRIPTION:
This study has three study visits: a consenting visit (~1 hour), a screening visit (~4 hours), and an ambulatory visit (~8 hours).

Visit 1: The participant will have the study explained to their satisfaction and sign the consent form, if the participant chooses to participate. A urine sample is collected to test for urinary tract infections and a prophylactic antibiotic is prescribed.

Note: The participant is asked to refrain from taking medications related to bladder relaxation (Ditropan, Oxybutynin, Detrol, Tolterodine Tartate, Tofranil, Imipramine, Urimax, Xanodine, Enablex, Darifenain) as these will interfere with the study. When to stop these medications will be discussed with the participant at this visit.

Visit 2: The participant will have a urodynamic screening visit to confirm NDO activity, determine the response to stimulation, and determine the most effective stimulation parameters for genital nerve stimulation.

* Urodynamics involves a catheter being inserted into the bladder to collect pressure readings from the bladder, and urethral sphincter, as well as infuse saline (salt water) into the bladder. This will be done up to 6 times, with and without stimulation, over the course of the 4 hour screening visit.
* During urodynamics a catheter is also inserted into the rectum. This sensor detects abdominal pressure during urodynamics and is used to determine the pressure in the bladder.

Note: There is an optional procedure that can be done in this visit called anorectal manometry (ARM). The rectal catheter that is inserted during urodynamics can also be used to investigate bowel function. If interested, the participant would be asked to perform several actions (cough, push as is if to defecate, or squeeze as if to withhold a bowel movement) and the response of the anal sphincter and rectum are measured.

Visit 3: If the participant has confirmed NDO, the participant will be invited to a longer visit (~8 hours) wherein the participant will test the full closed-loop stimulation system. The person will be asked to stay at the hospital for this visit but are encouraged to move about the building. This could involve going to the cafeteria or other public spaces. To accomplish closed-loop control of bladder function it will be necessary to:

* Insert a sensor into the bladder (UroMonitor) through the urethra. This sensor has been designed to stay inside the bladder and measure pressure without requiring a catheter to remain in the urethra. Once the study is completed the sensor will be retrieved via a suture that remains in the urethra.
* Confirm that the sensor is accurately detecting bladder pressure by comparing sensor values with urodynamics values. This will be done by using a urodynamics catheter and sensor at the same time for a short time.
* Having genital nerve stimulation electrodes affixed to the appropriate areas of the genitals. For men, these electrodes are put on the top of the penis. For women, these electrodes are placed on the labia majora near the clitoris. A ground electrode will be put on the inner thigh for both men and women. These electrodes will be connected to a transcutaneous electrical nerve stimulation (TENS) unit calibrated to deliver the appropriate current parameters for that participant (determined in visit 2).
* Donning the closed-loop system. The closed-loop system detects the sensor data, uses an algorithm to determine if stimulation should be applied, and then turns on the stimulation unit.

Once the participant is instrumented, the participant will be able to move about the building without restriction. This could include going to the cafeteria and moving through the hallways, rather than being sedentary in a procedure room. A study member will accompany the participant as the participant ambulates throughout the building and uses a computer tablet to view the bladder data.

Depending on how long it takes for the bladder to naturally fill, it may be possible to collect data from two fill-void cycles (~3 hours each). After data collection, the participant will be taken back to the procedure room and the instrumentation will be removed. That includes removal of the bladder sensor by the urologist on the study.

Participants will be asked for feedback which will include: what the participant experiences during the study, the design of the system, function of the system, any bladder related sensations, if the participant feels that the system would benefit quality of life, and if the participant would be likely to use the system.

ELIGIBILITY:
Inclusion Criteria:

* Suprasacral SCI (above L5/S1 level of the spinal cord)
* Neurologically stable
* Mature skeleton
* At least 6 months post-injury
* Neurogenic detrusor overactity (NDO) confirmed by urodynamic study

Exclusion Criteria:

* Active sepsis
* Open pressure ulcers on or around the pelvis (electrode sites)
* Significant trauma, erosion, or stricture of the urethra
* History of autonomic dysreflexia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
successful reduction of neurogenic bladder spasms | within 2 weeks of completing the screening visit
  The closed-loop system has been designed to detect neurogenic bladder spasms (contractions) and to turn on a device to deliver genital nerve stimulation. Genital nerve stimulation has been shown previously to relax NDO bladder spasms and therefore allow for increased capacity, longer time between catheterization, and a reduction in incontinence episodes. The outcome for this feasibility trial will be the ability of the system to perform within expected parameters (<5% false negative, <10% false positive, <5 s response time) to control NDO bladder contractions.

SECONDARY OUTCOMES:
Documentation of NDO with cystometrogram (urodynamics) | within 1 week of signing consent form
  To confirm the presence of NDO a cystometrogram will be conducted. This procedure uses a triple-lumen catheter inserted into the bladder which is used to fill the bladder with saline, measure bladder pressure, and measure urethral pressure. As the bladder is filled with saline the pressure readings will show if there are NDO contractions (sharp increase in bladder pressure AND an increase in sphincter pressure). This confirmation is necessary for eligibility in the study and can be informative for the participant.
Comparison of bladder activity with and without genital nerve stimulation | within 1 week of signing consent form
  During the screening visit (visit 2) the participant will undergo urodynamics testing to verify NDO. After verification of NDO, the procedure will be repeated with either effective or sham stimulation (up to 6 times total). This is to calibrate the stimulation parameters (amplitude) to ensure effective stimulation as well as to collect data regarding changes in bladder function due to genital nerve stimulation.

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Bourbeau, PhD, Principal Investigator — MetroHealth Rehabilitation Institute of Ohio
Locations (1):
- Metrohealth Medical System, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
There is no intention of sharing individual participant data with other researchers.